CLINICAL TRIAL: NCT04441892
Title: Phase II Novel Low Cost QTc Meter for Long QT Syndrome Screening in Primary Care
Brief Title: Low Cost QTc Meter for Long QT Syndrome Screening in Primary Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID, lack of funding and interruption of patient recruitment led to ending the study early.
Sponsor: Mayo Clinic (Other)
Collaborators: Blue Ox Healthcare Partners (Industry); Minnesota Health Solutions (Industry); iCardiac Technologies, Inc. (Industry)
Responsible Party: Principal Investigator, Michael J. Ackerman, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 18-006014
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Long QT Syndrome
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- QTc Meter (Experimental): Infants/Children (Day 0-Age 5) will participate in this study as minimal risk. Patients will record 30 seconds of data that is collected on the QTc Screening device
  Interventions: Device: QTc Meter
- QTc Meter - Healthy Controls (Experimental): Infants/Children (Day 0-Age 5) will participate in this study as minimal risk. Patients will record 30 seconds of data that is collected on the QTc Screening device.
  Interventions: Device: QTc Meter

INTERVENTIONS:
Device: QTc Meter — Development and evaluation of an inexpensive diagnostic device (the QTc Meter) to support simplified widespread screening in the primary care environment for both congenital long QT syndrome (LQTS) and acquired/drug induced-LQTS.

SUMMARY:
The purpose of this study is to further develop and evaluate a diagnostic procedure suitable for use in an inexpensive diagnostic instrument suitable for screening for Long QT Syndrome (LQTS) in the primary care environment.

DETAILED DESCRIPTION:
The study will involve acquiring ECG data in a cohort of up to 1,000 newborns and infants (500 controls (non-LQTS) and 500 LQTS newborns and infants) that are being seen in the Gonda SL ECG Lab (or Baldwin Building)and enrolled during their appointment for a clinically indicated 12-lead ECG. A second arm of Phase II of this study will include approaching 50 healthy subjects at the Baldwin Building to seek interest in participation which will consist of (1) 30 second device recording to help further calibrate and test the device for optimal enhancement. These 50 subjects will not be required to have a clinical or research 12-lead ECG as the investigators will be simply testing the efficiency and accuracy of the device. LQTS will be studied in order to assess the ability of the LQTS screener to accurately detect a patient with established QT prolongation in the context of distinct and varied T wave morphologies The advanced prototype will be placed in the same manner as the device used in Phase I of the study by being lightly placed on the child as pictured below. Similarly, the investigators will use ultrasound gel to obtain a better reading, if applicable. Once completed, a photograph of the torso of the child will be taken from the same views as before (one aerial view and one side view) with neither the head nor the face in the picture. Coded ECG-tracings will be transmitted to the app and shared with Blue Ox Health Corporation and Minnesota Health Solutions as done previously in phase I. Additionally, coded tracings and data from the 12-lead ECG will be shared with Blue Ox Health Corporation and Minnesota Health Solutions to aid in comparison to device tracings and optimization of the algorithm. The 12-lead ECG will be obtained from the subject's medical record and coded before being shared with collaborators. Study coordinators will also review the patient's medical record to determine whether the participants have been diagnosed with a genetic disease.

ELIGIBILITY:
Inclusion Criteria:

* Infants (Day 0 - 5 years).
* Long QT Syndrome(LQTS).
* Newborns without LQTS (Controls).
* Parental willingness to provide informed consent and follow the study protocol.

Exclusion Criteria:

* Children > 5 years old.
* Those with genetically elusive LQTS.
* Infants with congenital heart disease.
* Infants born < 32 weeks EGA.
* Patients with a cardiac device implant (pacemaker/ICD).

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ackerman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QTc Meter | QTc Meter - Healthy Controls
Started | 28 | 5
Completed | 28 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QTc Meter | QTc Meter - Healthy Controls | Total
Number analyzed (Participants) | 28 | 5 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.2 (1.5) | 2.8 (1.6) | 2.2 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 1 | 16
  Male | 13 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 27 | 4 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  White | 27 | 3 | 30
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 5 | 33

OUTCOME MEASURES:

1. Primary Outcome: Low Cost QTc Meter for Long QT Syndrome Screening
Description: Number of subjects to have a successful tracing recorded with the QTc Meter in Participants with or without Long QT Syndrome between the ages of 0 and 5
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | QTc Meter | QTc Meter - Healthy Controls
Number analyzed (Participants) | 28 | 5
Participants | 20 | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 1 day on all participants.
Arm/Group | QTc Meter | QTc Meter - Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/5
Other Adverse Events (participants affected / at risk) | 0/28 | 0/5

LIMITATIONS AND CAVEATS:
Last patient enrolled in February of 2020. Enrollment was paused because of stay-at-home COVID mandates and even when general clinical operations resumed, elective clinical studies like these were not immediately resumed in the ECG monitoring lab to limit the number of people around patients. By the time recruitment could resume, the collaborating company had run out of funding for the study and the study was terminated. Study only enrolled 33 participates out of anticipated 1050.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT04441892/Prot_000.pdf